CLINICAL TRIAL: NCT01362075
Title: Pain Management After Shoulder Arthroplasty: A Randomised Clinical Trial of Interscalene Block and Local Infiltration Analgesia
Brief Title: Pain Management After Shoulder Prosthesis: A Clinical Trial of Nerve Block and Local Infiltration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After 3 years of recruitment, the study was stopped due to time constraints.
Sponsor: Horsens Hospital (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other); The Hede Nielsen Family Foundation (Other); Central Denmark Region (Other); The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Karen Toftdahl Bjørnholdt, MD, Horsens Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTB-001; M-20110084 (Other: Central Denmark Region Ethics Committee)
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Pain, Postoperative
Keywords: Shoulder Arthroplasty; Local infiltration analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local infiltration analgesia (Experimental)
  Interventions: Procedure: Local infiltration analgesia
- Interscalene catheter (Active Comparator)
  Interventions: Procedure: Interscalene catheter

INTERVENTIONS:
Procedure: Local infiltration analgesia — 150 ml ropivacaine, of which 100 ml is with adrenalin
  Other Names: LIA
  Arms: Local infiltration analgesia
Procedure: Interscalene catheter — 7 ml ropivacaine interscalene block via catheter, subsequently given 5 ml/h and possibility of 5 ml bolus for the first 48 hours.
  Other Names: interscalene block
  Arms: Interscalene catheter

SUMMARY:
The purpose of this study is to determine the efficacy of local infiltration analgesia as compared to 48-hour interscalene block in treating pain after shoulder arthroplasty. The investigators hypothesize a reduced pain score and use of supplemental analgesic medication during the first three postoperative days using local infiltration analgesia.

ELIGIBILITY:
Inclusion Criteria:

* elective primary shoulder arthroplasty

Exclusion Criteria:

* reverse or delta prosthesis
* recent fracture near the shoulder
* allergic to amid-type local analgesics
* operation not under general anaesthesia
* incompetent, pregnant, below 18 or above 90 years old
* severe chronic neurogenic pain or sensory disturbances in the shoulder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Supplemental analgesics ingested | First 24 hours postoperatively

SECONDARY OUTCOMES:
Pain score | First 72 hours postoperatively
Supplemental analgesics ingested | First 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Bjørnholdt, MD, Principal Investigator — Horsens Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus Hospital, Aarhus, Denmark
  - Horsens Hospital, Horsens, Denmark